CLINICAL TRIAL: NCT01986855
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Ertugliflozin (MK-8835/PF-04971729) in Subjects With Type 2 Diabetes Mellitus With Stage 3 Chronic Kidney Disease Who Have Inadequate Glycemic Control on Background Antihyperglycemic Therapy
Brief Title: A Study of the Efficacy and Safety of Ertugliflozin in Participants With Type 2 Diabetes Mellitus With Stage 3 Chronic Kidney Disease Who Have Inadequate Glycemic Control on Antihyperglycemic Therapy (MK-8835-001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-001; 2013-003587-31 (EudraCT Number); B1521016 (Other: Pfizer)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ertugliflozin (5 mg) (Experimental): Ertugliflozin, 5 mg, oral, one 5 mg ertugliflozin tablet and one placebo tablet, once daily for 52 weeks
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo 10 mg
- Ertugliflozin (15 mg) (Experimental): Ertugliflozin, 15 mg, oral, one 5 mg and one 10 mg tablet, once daily for 52 weeks
  Interventions: Drug: Ertugliflozin 10 mg
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo 5 mg; Drug: Placebo 10 mg

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin, oral, 5 mg tablet once daily for 52 weeks
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin (5 mg)
Drug: Placebo 5 mg — Placebo to ertugliflozin, oral, tablet, 5 mg tablet once daily for 52 weeks
  Arms: Placebo
Drug: Ertugliflozin 10 mg — Ertugliflozin, oral, tablet, 10 mg tablet once daily for 52 weeks
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin (15 mg)
Drug: Placebo 10 mg — Placebo to ertugliflozin, oral, tablet, 10 mg tablet once daily for 52 weeks
  Arms: Ertugliflozin (5 mg); Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ertugliflozin (MK-8835/PF-04971729) in participants with Type 2 diabetes mellitus with Stage 3 Chronic Kidney Disease (CKD) who have inadequate glycemic control on background antihyperglycemic therapy. The duration of this trial will be up to 67 weeks. This study will consist of a 1-week Screening Period, a 10-week wash-off period from metformin, if needed, and a 2-week placebo run-in period, a 52-week double-blind treatment period, and a 14-day post-treatment follow-up period. The primary objective of this trial is to assess the hemoglobin A1C (A1C)-lowering efficacy of the addition of ertugliflozin compared to the addition of placebo with an underlying hypothesis that addition of treatment with ertugliflozin provides greater reduction in A1C compared to the addition of placebo; the primary objective will be tested for both 5-mg and 15-mg doses of ertugliflozin.

DETAILED DESCRIPTION:
Participants who meet protocol-defined glycemic rescue criteria will be permitted to have an adjustment in the dose(s) of background antihyperglycemic agent (AHA) therapy or addition of new AHA therapy as directed by their investigator until the participant no longer meets the rescue criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes mellitus in accordance with American Diabetes Association guidelines
* Have Stage 3 chronic kidney disease
* On stable diabetes therapy (diet/exercise therapy alone or anti-hyperglycemic agents [AHA] monotherapy or combination therapy) for at least 6 weeks prior to study participation OR on metformin (with or without diet/exercise therapy or other AHA therapy) and is willing to undergo a 10-week metformin wash-off period
* Have an estimated glomerular filtration rate (eGFR) of ≥30 to <60 mL/min/1.73m^2
* Body Mass Index (BMI) greater than or equal to 18.0 kg/m^2
* Male, postmenopausal female or surgically sterile female
* If a female of reproductive potential, agrees to remain abstinent or to use (or have their partner use) 2 acceptable combinations of birth control while participating in the trial and for 14 days after the last use of study drug.

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrine disorders, drug - or chemical-induced, and post-organ transplant)
* History of nephrotic range proteinuria with hypoalbuminemia and edema
* History of rapidly progressive glomerulonephritis, lupus nephritis, renal or systemic vasculitis, renal artery stenosis with renovascular hypertension, or ischemic nephropathy
* History of familial renal glucosuria
* History of renal dialysis or renal transplant or renal disease requiring treatment with any immunosuppressive agent
* A known hypersensitivity or intolerance to any (sodium-glucose co-transporter 2) SGLT2 inhibitor
* On a weight-loss program or weight-loss medication or other medication associated with weight changes and is not weight stable
* Has undergone bariatric surgery within the past 12 months
* Has been treated with rosiglitazone or other SGLT2 inhibitors within 12 weeks of study participation
* Has active, obstructive uropathy or indwelling urinary catheter
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study participation
* A history of malignancy ≤5 years prior to study participation, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* Known history of Human Immunodeficiency Virus (HIV)
* Has blood dyscrasias or any disorders causing hemolysis or unstable red blood cells or any other clinically significant hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* A medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease
* Has any clinically significant malabsorption condition
* If taking thyroid replacement therapy, has not been on a stable dose for at least 6 weeks prior to study participation
* Has been previously randomized in a study with ertugliflozin
* Has participated in other studies involving an investigational drug within 30 days prior or during study participation
* Has undergone a surgical procedure within 6 weeks prior to or during study participation
* Has a positive urine pregnancy test
* Is pregnant or breast-feeding, or is planning to conceive during the trial, including 14 days following the last dose of study medication
* Planning to undergo hormonal therapy in preparation to donate eggs during the trial, including 14 days following the last dose of study medication
* Excessive consumption of alcoholic beverages or binge drinking
* Has donated blood or blood products within 6 weeks of study participation or plans to donate blood or blood products at any time during the trial

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Grunberger G, Camp S, Johnson J, Huyck S, Terra SG, Mancuso JP, Jiang ZW, Golm G, Engel SS, Lauring B. Ertugliflozin in Patients with Stage 3 Chronic Kidney Disease and Type 2 Diabetes Mellitus: The VERTIS RENAL Randomized Study. Diabetes Ther. 2018 Feb;9(1):49-66. doi: 10.1007/s13300-017-0337-5. Epub 2017 Nov 20. PMID 29159457
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 13 countries, including 171 trial centers; 1709 participants were screened and 468 were randomized.
Pre-assignment Details: Eligible participants began a ≥10-week metformin wash-off during which participant's antihyperglycemic agents (AHAs) could be adjusted.
  All participants entered a 2-week placebo run-in period.
Groups:
- Ertugliflozin 5 mg: Ertugliflozin, oral, 5-mg tablet once daily for 52 weeks. Participants also received a 10-mg matching placebo tablet once daily for 52 weeks.
- Ertugliflozin 15 mg: Ertugliflozin, oral, 5-mg and 10-mg tablet once daily for 52 weeks
- Placebo: Placebo, oral, tablet, 5-mg or 5-mg and 10-mg tablet once daily for 52 weeks
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Started | 158 | 156 | 154
Treated | 158 | 155 | 154
Completed | 145 | 142 | 143
Not Completed | 13 | 14 | 11
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 3 | 4 | 4
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Screen Failure | 0 | 1 | 0
Not completed — Participant Moved | 0 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 8 | 5

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants was the All-Participants-As-Treated population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo | Total
Number analyzed (Participants) | 158 | 155 | 154 | 467
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (8.3) | 67.5 (8.5) | 67.5 (8.9) | 67.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 80 | 82 | 236
  Male | 84 | 75 | 72 | 231
Baseline Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percentage] — Population: Participants with baseline data for A1C.
  Percentage
    number analyzed (Participants) | 154 | 151 | 152 | 457
    (all) | 8.20 (1.02) | 8.17 (0.87) | 8.08 (0.89) | 8.15 (0.93)
Baseline Weight [Mean (Standard Deviation); unit: Kilograms] | 89.4 (22.5) | 85.8 (17.4) | 90.4 (18.9) | 88.5 (19.8)
Baseline Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: Participants with baseline data for FPG.
  mg/dL
    number analyzed (Participants) | 157 | 155 | 154 | 466
    (all) | 160.9 (56.4) | 157.5 (47.8) | 156.9 (56.4) | 158.5 (53.6)
Baseline Estimated glomerular filtration rate (eGFR) [Number; unit: Participants] — Stratification Factor: eGFR (mL/min/1.73m^2)
  Participants
    ≥30 to <45 | 52 | 53 | 54 | 159
    ≥45 to <60 | 106 | 102 | 100 | 308
Stratification Factor: Insulin at randomization [Number; unit: Participants] — Insulin at randomization? (Yes/No)
  Participants
    No | 69 | 68 | 66 | 203
    Yes | 89 | 87 | 88 | 264

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 26 - Excluding Rescue Approach
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 26 A1C minus the Week 0 A1C. Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants who took at least 1 dose of study treatment and had at least 1 assessment at or after baseline for the change from baseline at Week 26 A1C endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 154
Percentage | -0.29 [-0.44 to -0.14] | -0.41 [-0.56 to -0.27] | -0.26 [-0.41 to -0.11]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.807, Constrained longitudinal data analysis — The cLDA model included fixed effects for treatment, time, eGFR stratum (<45 or ≥45 mL/min/1.73m^2), baseline treatment with insulin stratum (yes/no), and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.03, 95% CI 2-sided [-0.23 to 0.18]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.155, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in the least squares means = -0.15, 95% CI 2-sided [-0.35 to 0.06]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 54 weeks
Population: The analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 154
Percentage of participants | 84.8 | 74.2 | 81.2
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in Percentages vs. Placebo = 3.6, 95% CI 2-sided [-4.8 to 12.1] — Miettinen & Nurminen Method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in Percentages vs. Placebo = -7.0, 95% CI 2-sided [-16.3 to 2.3] — Miettinen & Nurminen Method

3. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: The analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 154
Percentage of participants | 8.2 | 3.9 | 5.2
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; Difference in Percentages vs. Placebo = 3.0, 95% CI 2-sided [-2.7 to 9.0] — Miettinen & Nurminen Method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; Difference in Percentages vs. Placebo = -1.3, 95% CI 2-sided [-6.5 to 3.7] — Miettinen & Nurminen Method

4. Secondary Outcome: Change From Baseline in A1C at Week 26 - Baseline eGFR ≥45 to <60 mL/Min/1.73m^2 Stratum - Excluding Rescue Approach
Description: as for outcome 1
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants with a Baseline eGFR of ≥45 to <60 mL/min/1.73m^2 and who took at least 1 dose of study treatment and had at least 1 assessment at or after baseline for the change from baseline at Week 26 A1C endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 105 | 97 | 99
Percentage | -0.31 [-0.49 to -0.13] | -0.37 [-0.56 to -0.18] | -0.28 [-0.47 to -0.08]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.828, Constrained longitudinal data analysis — The cLDA model included fixed effects for treatment, time, baseline treatment with insulin stratum (yes/no), and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.03, 95% CI 2-sided [-0.28 to 0.23]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.496, Constrained longitudinal data analysis — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -0.09, 95% CI 2-sided [-0.35 to 0.17]

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26 - Baseline eGFR ≥45 to <60 mL/Min/1.73m^2 Stratum - Excluding Rescue Approach
Description: This change from baseline reflects the Week 26 body weight minus the Week 0 body weight. Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants with a Baseline eGFR of ≥45 to <60 mL/min/1.73m^2 and who took at least 1 dose of study treatment and had at least 1 assessment at or after baseline for the change from baseline at Week 26 body weight endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 105 | 97 | 99
Kilograms | -1.31 [-1.86 to -0.76] | -1.39 [-1.97 to -0.81] | 0.46 [-0.13 to 1.04]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — The cLDA model included fixed effects for treatment, time, baseline treatment with insulin stratum (yes/no), and the interaction of time by treatment. Time was treated as a categorical variable. P-value is nominal; Difference in the least squares means = -1.77, 95% CI 2-sided [-2.57 to -0.96]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 5, analysis 1]; Difference in the least squares means = -1.84, 95% CI 2-sided [-2.66 to -1.02]

6. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26 - Baseline eGFR ≥45 to <60 mL/Min/1.73m^2 Stratum - Excluding Rescue Approach
Description: This change from baseline reflects the Week 26 sitting systolic blood pressure minus the Week 0 sitting systolic blood pressure. Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants with a Baseline eGFR of ≥45 to <60 mL/min/1.73m^2 and who took at least 1 dose of study treatment and had at least 1 assessment at or after baseline for the change from baseline at Week 26 sitting systolic blood pressure endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 105 | 97 | 99
mmHg | -2.33 [-4.98 to 0.33] | -4.36 [-7.11 to -1.62] | -0.90 [-3.73 to 1.92]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.451, Constrained longitudinal data analysis — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -1.42, 95% CI 2-sided [-5.13 to 2.29]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.072, Constrained longitudinal data analysis — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -3.46, 95% CI 2-sided [-7.24 to 0.31]

7. Secondary Outcome: Change From Baseline in FPG at Week 26 - Baseline eGFR ≥45 to <60 mL/Min/1.73m^2 Stratum - Excluding Rescue Approach
Description: This change from baseline reflects the Week 26 FPG minus the Week 0 FPG. Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants with a Baseline eGFR ≥45 to <60 mL/min/1.73m^2 and who took at least 1 dose of study treatment and had at least 1 assessment at or after baseline for the change from baseline at Week 26 FPG endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 105 | 97 | 99
mg/dL | -11.76 [-21.07 to -2.45] | -20.47 [-30.20 to -10.73] | -4.95 [-15.03 to 5.13]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.291, Constrained longitudinal data analysis — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -6.81, 96% CI 2-sided [-19.47 to 5.85]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.019, Constrained longitudinal data analysis — [p-value comment as in outcome 5, analysis 1]; Difference in the least squares means = -15.51, 95% CI 2-sided [-28.50 to -2.53]

8. Secondary Outcome: Percentage of Participants With A1C <7.0% (<53 mmol/Mol) at Week 26 - Baseline eGFR ≥45 to <60 mL/Min/1.73m^2 Stratum - Excluding Rescue Approach
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Week 26
Population: The analysis population included all randomized participants with a Baseline eGFR ≥45 to <60 mL/min/1.73m^2 and who took at least 1 dose of study treatment and had at least 1 assessment at Week 26 for the percentage of participants with an A1C <7% at Week 26 endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 105 | 97 | 99
Percentage of participants | 16.2 | 11.3 | 12.1
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.713, Logistic regression model — Adjusted Odds Ratio based on a logistic regression model fitted with fixed effects for treatment, baseline treatment with insulin stratum (yes/no), and a covariate for baseline A1C; Adjusted Odds Ratio = 1.16, 95% CI 2-sided [0.53 to 2.56]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.890, Logistic regression model — [p-value comment as in outcome 8, analysis 1]; Adjusted Odds Ratio = 1.06, 95% CI 2-sided [0.44 to 2.55]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Arm/Group | Placebo | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Serious Adverse Events (participants affected / at risk) | 24/154 | 26/158 | 30/155
Other Adverse Events (participants affected / at risk) | 68/154 | 82/158 | 62/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | Ertugliflozin 5 mg (N=158) | Ertugliflozin 15 mg (N=155)
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (7)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sciatic nerve palsy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | Ertugliflozin 5 mg (N=158) | Ertugliflozin 15 mg (N=155)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 10 (10) | 4 (4)
Bronchitis (Infections and infestations) | 6 (7) | 8 (8) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (8) | 9 (10) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 9 (9) | 11 (12)
Urinary tract infection (Infections and infestations) | 15 (20) | 9 (11) | 12 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 45 (216) | 49 (423) | 32 (281)
Dizziness (Nervous system disorders) | 1 (1) | 9 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) | 3 (3)

LIMITATIONS AND CAVEATS:
After unblinding, analysis of retained plasma samples revealed unreported metformin use by ~17% of participants. Neither dose nor frequency of the protocol-prohibited metformin use is known. This potentially confounds glycemic analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.